CLINICAL TRIAL: NCT05393700
Title: Effects of Early Sleep After Action Observation Therapy on Balance in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Principal Investigator, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLF22/01
Record Dates: First submitted 2022-05-20; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Old Age; Debility; Balance; Distorted
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AOT-sleep (Experimental): They will be asked to watch video-clips representing motor contents before sleeping.
  Interventions: Behavioral: Action Observation Therapy
- AOT-control (Active Comparator): They will be asked to watch video-clips representing motor contents at least 12 hours before sleeping.
  Interventions: Behavioral: Action Observation Therapy
- Control (Sham Comparator): They will be asked to watch video-clips representing landscapes before sleeping.
  Interventions: Behavioral: Action Observation Therapy

INTERVENTIONS:
Behavioral: Action Observation Therapy — Action Observation Therapy implies the observation of video-clips representing motor tasks alone or followed by imagination and/or imitation of observed tasks.

SUMMARY:
The study aims at investigating the effects of an early sleep window after Action Observation Therapy (AOT) on balance in elderly. Forty-five healthy-like elderly will be enrolled and randomized into 3 groups (AOT-sleep, AOT-control and Control) performing a 3-week AOT. AOT-sleep and AOT-control will be asked to watch video-clips showing motor contents before sleeping or at least 12 hours before sleeping, respectively, whereas Control will be asked to watch landascape video-clips before sleeping. Participants will be assessed before and after training and at 1 month follow-up for balance outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk for at least 100 meters with no assistance or aids

Exclusion Criteria:

* Musculoskeletal disorders able to affect balance
* Traumas and/or injuries and/or surgery at the level of the lower limbs, spine in the previous year
* Sleep disorders
* Drugs able to affect sleep
* Dementia or cognitive decline (MCI)
* Psychiatric or neurological disorders

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Lower Quarter Y-Balance Test | At baseline, 3 weeks and 1 month after the training end
  The outcome measure is aimed at investigating changes in terms of static balance
Changes in 10-Meter Walking Test | At baseline, 3 weeks of training and 1 month after the training end
  The outcome measure is aimed at investigating changes in terms of gait speed
Changes in Timed Up and Go Test | At baseline, 3 weeks of training and 1 month after the training end
  The outcome measure is aimed at investigating changes in terms of mobility
Changes in Four Step Square Test | At baseline, 3 weeks of training and 1 month after the training end
  The outcome measure is aimed at investigating changes in terms of dynamic balance

SECONDARY OUTCOMES:
Changes in center of pressure parameters | At baseline, 3 weeks of training and 1 month after the training end
  The outcome measure is aimed at investigating changes in terms of postural stability
Changes in Fall Efficacy Scale | At baseline, 3 weeks of training and 1 month after the training end
  The outcome measure is aimed at investigating changes in terms of fear of falling
Pittsburg Quality Sleep Index | 3 weeks
  The outcome measure is aimed at investigating the sleep quality in the training period. The scale ranges from 0 (better outcome) to 21 points (worse outcome)
Kinesthetic and Visual Imagery Questionnaire | At baseline
  The outcome measure is aimed at investigating the imagination ability of participants. The scale range from 0 (worse score) to 50 (better score).
Morningness Eveningness Scale | At baseline
  The outcome measure is aimed at investigating the chronotype of participants. The score ranges from 16 to 86 points. A score lower than 41 points indicates "evening types.", scores of 59 and above indicate "morning types", while scores between 42-58 indicate "intermediate types."
Euro Quality of Life - 5 dimensions | At baseline
  The outcome measure is aimed at investigating the quality of life of participants. The scale ranges from 0 (worse outcome) to 1 (better outcome).

IPD SHARING:
Plan to Share IPD: No